CLINICAL TRIAL: NCT07118501
Title: A Prospective, Post-Market, Clinical Follow-up Study of the Incompass™ Total Ankle System
Status: Not yet recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: FA-02-2024
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Arthritis; Osteoarthritis; Total Ankle Replacement; Total Ankle Prosthesis
Keywords: Total Ankle Replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Incompass™ Total Ankle System: Primary Total Ankle Replacement using the Incompass™ Total Ankle System
  Interventions: Device: Total Ankle Replacement

INTERVENTIONS:
Device: Total Ankle Replacement — Incompass™ Total Ankle System

SUMMARY:
The goal of this study is to demonstrate the safety and performance of the Incompass™ Total Ankle System after surgery over the standard follow-up period. The study will measure improvements in patient-reported information related to quality of life and pain following surgery. In order to do this, medical imaging (i.e. X-Rays, CT scans) which have been taken as part of routine care, will be reviewed. Any additional X-Rays conducted during the period of the research will also be reviewed.

The Incompass™ Total Ankle System has been cleared by the Food and Drug Administration (FDA). The products are already in use routinely in ankle replacement surgeries. No part of this study is experimental.

DETAILED DESCRIPTION:
It is anticipated that a total of 200 subjects will be enrolled at up to ten sites over a three year enrollment period. The study has been designed to follow the surgeon's standard of care for subjects treated with a total ankle replacement including imaging (x-rays and or CT scans).

The primary endpoint of this study is the 24-month total Ankle Osteoarthritis Scale (AOS) score improvement after index surgery (or Initial Assessment). Secondary endpoints include safety (adverse events, reoperation, and survivorship) as well as performance measures (radiographic assessments, PROMIS Global Health questionnaire, Foot and Ankle Ability Measure [FAAM] and Total Ankle Replacement [TAR] Satisfaction questionnaires).

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be willing and able to sign a written approved informed consent form (ICF) approved by Institutional Review Board (IRB) or Ethics Committee (EC)
2. Participants must be males or non-pregnant females aged 21 years or older at the time of surgery;
3. Willing and able to comply with the requirements of the clinical investigation plan (CIP), including attend all required study visits.
4. The participant must be able to follow instructions and deemed capable of completing clinical investigation questionnaires.
5. Considered a candidate for total ankle replacement with the Incompass Total Ankle System in accordance with its legally approved Indication for Use (IFU).

Exclusion Criteria:

1. Participant with an ankle condition, as determined by the investigator, to be an inappropriate candidate for total ankle replacement;
2. Participant is currently enrolled in or plans to enroll in any concurrent drug and/or device clinical investigation that, in the opinion of the Investigator, may confound results;
3. Any participant that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.44.
4. Participants who have participated previously in this clinical trial and who have been withdrawn.
5. Participant who is, or will be, inaccessible for follow-up
6. Participant is pregnant or intends to become pregnant during the course of the study.
7. Participants with a medical or physical condition that, in the opinion of the Investigator, would preclude safe participation in the clinical investigation.
8. Participants requiring revision total ankle replacement of the ankle being considered for the study;
9. Participants with a failed previous ankle surgery (e.g., takedown fusion)
10. Participants with any infection at the ankle site or infections at distant sites that could migrate to the ankle, including sepsis and osteomyelitis;
11. Participants with compromised vascularity that would inhibit blood supply to the operative site;
12. Neuropathic arthropathy of the joint;
13. Insufficient bone stock or bone quality that cannot provide adequate support of the device;
14. Participants who have documented or suspected sensitivity to the implant materials.
15. Participants with inadequate neuromuscular status or those having poor skin coverage around the joint, which would make the procedure unjustifiable
16. Participant who routinely place excessive loads on their ankle as caused by activity and/or patient weight, per investigator discretion; or
17. Any mental or neuromuscular disorder that would create an unacceptable risk of failure or complications in postoperative care.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No specific methods (such as randomization, blinding or stratification) for assigning participants are used in this protocol. Consecutive participants at each site meeting all of the eligibility criteria will be considered for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2038-09-01 (Estimated)

PRIMARY OUTCOMES:
Ankle Osteoarthritis Scale (AOS) | Baseline, 6 month, 1 Year, 2 Year, 5 Year, 7 Year, 10 Year
  The AOS questionnaire consists of two 9-item subscales: one for pain and one for disability. Each subscale uses a visual analogue scale where patients mark a point on a 100mm horizontal line anchored by "No pain" and "Worst pain imaginable" for pain, or "No difficulty" and "So difficult unable" for disability

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | Baseline, 6 month, 1 Year, 2 Year, 5 Year, 7 Year, 10 Year
  The FAAM has 29 questions and two components that are scored independently: an Activities of Daily Living (ADL) subscale and a Sports subscale. Each subscale is scored from 0 to 100 points, with higher scores representing better function.
PROMIS Scale v1.2- Global Physical Health Score | Baseline, 6 Month, 1 Year, 2 year, 5 Year, 7 year, 10 Year
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score." The average "TScore" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
PROMIS Scale v1.2- Global Mental Health Score | Baseline, 6 Month, 1 Year, 2 year, 5 Year, 7 year, 10 Year
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score." The average "TScore" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
TAR Satisfaction | 6 month, 1 Year, 2 Year, 5 Year, 7 Year, 10 Year
  Patient satisfaction with the Incompass™ Total Ankle System post-operatively is assessed utilizing a four-point scale: excellent, good, fair and poor.
Radiographic Findings | Baseline, 6 months, 1 year, 2 year, 5 year, 7 year, 10 year.
  Radiographic assessment for component loosening and/or subsidence, any osteolysis and/or cyst formation early and through the lifetime of the implant.
Safety - Adverse Event | Baseline to 10 years postoperative
  The incidence of device-related Adverse Events by 10 years, as collected and reported by the Investigator
Safety - Survivorship | Baseline to 10 years.
  The survivorship rate by 10 years, as defined with a Kaplan-Meier survivorship analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities

IPD SHARING:
Plan to Share IPD: No